CLINICAL TRIAL: NCT06998017
Title: The Feasibility of Low-Volume High Intensity Interval Training on Inpatient Stroke Rehab
Brief Title: The Feasibility of LVHIIT on Inpatient Stroke Rehab
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00160192
Record Dates: First submitted 2025-03-05; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Stroke; High Intensity Interval Training; Aerobic Fitness; Physical Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Volume High Intensity Interval Training (Experimental): This is the only arm in the study as it is a feasibility trial.
  Interventions: Other: Low Volume High Intensity Interval Training

INTERVENTIONS:
Other: Low Volume High Intensity Interval Training — Participants will conduct aerobic exercise on a total body recumbent stepper to get their heart rates to levels consistent with high intensity exercise.

SUMMARY:
The objective of this study is to explore the safety and feasibility of conducting low-volume, high-intensity interval training (HIIT) on a total body recumbent stepper (TBRS) in persons with stroke in an inpatient rehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

* -Both sexes between the age of 18-85 years at time of consent
* Ischemic or hemorrhagic stroke at consent. People with stroke and newly diagnosed cardiovascular complications had >50% prevalence of recurrent stroke at 5 years. Index stroke or recurrent stroke on same side as index stroke will be allowed.
* Exercise continuously for minimum of 30 watts for 3 minutes on the recumbent stepper to demonstrate ability to perform the exercise test or therapist confirmation/documentation of participant's ability to use the recumbent stepper.
* No aerobic exercise contraindications or other safety/physical concerns during the submaximal exercise test determined by the therapy team or inpatient physicians.
* Able to communicate with investigators, follow 2-step command & correctly answer consent comprehension questions

Exclusion Criteria:

* Implanted pacemaker or defibrillator limiting exercise performance
* Reported pain that limits or interferes with activities of daily living and physical activity/exercise
* Acute Myocardial Infarction in the last 2 days
* Ongoing unstable Angina
* Active Endocarditis
* Symptomatic Severe Aortic Stenosis
* Decompensated Heart Failure
* Acute Pulmonary Embolism, Pulmonary Insufficiency, or Deep Veinous Thrombosis
* Acute Myocarditis or Pericarditis
* Other significant neurologic, orthopedic, or peripheral vascular conditions that would limit exercise participation
* Oxygen-dependent chronic obstructive pulmonary disease
* Neurological disease (Multiple Sclerosis, Alzheimer's disease, Parkinson's disease)
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Safety of LVHIIT (low volume high intensity interval training) on total body recumbent stepper | 2-3 months
  Treatment related adverse events will be defined as the presence of study-related cardiac or serious adverse events. The Investigators hypothesize that low-volume, short-interval, TBRS HIIT will have no incidents of treatment related adverse events in participants with subacute stroke while admitted to inpatient rehabilitation during HIIT (H1a) and within the 30 minutes following HIIT cessation (H1b).
Adherence of LVHIIT (low volume high intensity interval training) on total body recumbent stepper | 2-3 months
  Feasibility will be assessed by adherence to the exercise session, attainment of target heart rates, and acceptability of the exercise. Adherence will measured by ≥ 75% of participants complete the entire 10-minute HIIT bout (H2a). Units will be the number of participants that are able to finish the full 10 minute bout of exercise.
Attainment of LVHIIT (low volume high intensity interval training) on total body recumbent stepper | 2-3 months
  Feasibility will be assessed by adherence to the exercise session, attainment of target heart rates, and acceptability of the exercise. Attainment will be measured by ≥75% of participants will reach target heart rates (75%-85% max HR) during ≥75% of the high-intensity intervals (H2b). Heart rates will be measured in beats per minute. HR max will be calculated using an algorithm that adjusts for age, or beta blocker use. Units will be the number of participants reaching target HR.
Acceptability of LVHIIT (low volume high intensity interval training) on total body recumbent stepper | 2-3 months
  Feasibility will be assessed by adherence to the exercise session, attainment of target heart rates, and acceptability of the exercise. To examine acceptability, the valid and reliable 8-item Physical Activity Enjoyment Scale (PACES-8) will be used, where higher scores indicate greater exercise enjoyment (H2c).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Arickx, MD, Principal Investigator — University of Kansas

DOCUMENTS (2):
  • Study Protocol (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT06998017/Prot_000.pdf
  • Informed Consent Form (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT06998017/ICF_001.pdf